CLINICAL TRIAL: NCT06922552
Title: Clinical Performance of Giomer Preceded by Etching Versus Resin-Based Sealants Applied on Permanent Molars Affected by Molar-Incisor Hypo-mineralization: A Randomized Clinical Trial
Brief Title: Clinical Performance of Giomer Preceded by Etching Versus Resin-Based Sealants Applied on Permanent Molars Affected by Molar-Incisor Hypo-mineralization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nayera Mohammed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Faculty of Dentistry Cairo Uni
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Molar Incisor Hypomineralization
Keywords: MIH; Giomer based sealants; Molar Incisor hypomineralization; Sealants; Rein based sealants
MeSH Terms: conditions — Molar Hypomineralization | interventions — Pit and Fissure Sealants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple (Participants, Care Provider, Outcome Assessor )
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Giomer based sealant applied on Permanent Molars Affected by MIH (Experimental): * Cleaning with a bristle brush and a non-fluoridated paste will be operated by a slow speed handpiece and absolute isolation (using rubber dam and Young's bow).
  * Phosphoric acid etch will be applied to the occlusal fissures for 30 seconds. Teeth will be washed using air-water spray for 30 seconds then drying using air for 15 seconds. Proper etching will be confirmed by a dull frosty-white appearance of the enamel An adequate amount of primer will be dispensed on the enamel surface of the pit and fissure using a brush then will be left undisturbed for 5sec. Gentle air blow for 3 sec and then dryness with stronger stream of air until a thin and uniform bonding layer is obtained.
  * The giomer sealant (BeautiSealant, Shofu, Kyoto, Japan) will be applied into the occlusal fissures applied Using the syringe needle tip and a brush into the pits and fissures. Stirring the sealant with the syringe-tip during or after placement will help eliminate any possible bubbles and enhance the fl
  Interventions: Procedure: Giomer pit and fissure sealant with etching applied on Permanent Molars Affected by MIH
- Resin based sealant applied on permanent molars affected by MIH (Active Comparator): * Cleaning with a bristle brush and a non-fluoridated paste will be operated by a slow speed handpiece and absolute isolation (using rubber dam and Young's bow).
  * Phosphoric acid etch will be applied to the occlusal fissures for 30 seconds. Teeth will be washed using air-water spray for 30 seconds then drying using air for 15 seconds. Proper etching will be confirmed by a dull frosty-white appearance of the enamel
  * The resin sealant will be applied Using the syringe needle tip and a brush into the pits and fissures. Stirring the sealant with the syringe-tip during or after placement will help eliminate any possible bubbles and enhance the flow into the pit and fissures. Photo - curing for the sealant will be done for 20 seconds using LED light curing unit. The tip of the light will be held as close as possible to the sealant, without actually touching the sealant.
  Interventions: Procedure: Resin based sealant applied on Permanent Molars Affected by MIH

INTERVENTIONS:
Procedure: Giomer pit and fissure sealant with etching applied on Permanent Molars Affected by MIH — * Cleaning with a bristle brush and a non-fluoridated paste will be operated by a slow speed handpiece and absolute isolation (using rubber dam and Young's bow).
  * Phosphoric acid etch will be applied to the occlusal fissures for 30 seconds. Teeth will be washed using air-water spray for 30 seconds then drying using air for 15 seconds. Proper etching will be confirmed by a dull frosty-white appearance of the enamel An adequate amount of primer will be dispensed on the enamel surface of the pit and fissure using a brush then will be left undisturbed for 5sec. Gentle air blow for 3 sec and then dryness with stronger stream of air until a thin and uniform bonding layer is obtained.
  * The giomer sealant (BeautiSealant, Shofu, Kyoto, Japan) will be applied into the occlusal fissures applied Using the syringe needle tip and a brush into the pits and fissures. Stirring the sealant with the syringe-tip during or after placement will help eliminate any possible bubbles and enhance the flow.
  Arms: Giomer based sealant applied on Permanent Molars Affected by MIH
Procedure: Resin based sealant applied on Permanent Molars Affected by MIH — Cleaning with a bristle brush and a non-fluoridated paste will be operated by a slow speed handpiece and absolute isolation (using rubber dam and Young's bow).
  * Phosphoric acid etch will be applied to the occlusal fissures for 30 seconds. Teeth will be washed using air-water spray for 30 seconds then drying using air for 15 seconds. Proper etching will be confirmed by a dull frosty-white appearance of the enamel
  * The resin sealant (UltraSeal XT™ hydro™) will be applied Using the syringe needle tip and a brush into the pits and fissures. Stirring the sealant with the syringe-tip during or after placement will help eliminate any possible bubbles and enhance the flow into the pit and fissures. Photo - curing for the sealant will be done for 20 seconds using LED light curing unit. The tip of the light will be held as close as possible to the sealant, without actually touching the sealant.
  the surfaces will be checked with an explorer to ensure that no voids were present.
  Arms: Resin based sealant applied on permanent molars affected by MIH

SUMMARY:
The goal of the study is to evaluate the clinical performance of giomer sealant preceded by etching versus resin-based sealants applied on first permanent molars affected by molar incisor hypomineralization (MIH)

The main question it aims to answer is :

Will the use of Giomer (Beautisealant, Shofu, Kyoto, Japan) Preceded by Etching result in similar clinical performance as Resin-Based Sealants(UltraSeal XT™ Plus™ by Ultradent) Applied on Permanent Molars Affected by Molar-Incisor Hypomineralization?

DETAILED DESCRIPTION:
Molar Incisor Hypomineralization (MIH) is a developmental defect impacting first permanent molars and incisors, characterized by enamel opacities, and reduced mineral content. This condition can cause aesthetic, functional, psychological, and behavioral problems in children. Moreover, there are dental treatment challenges associated with (MIH)which include behavior management, difficulty with local anesthesia, tooth hypersensitivity, and issues with restoration retention.

Teeth affected by (MIH) are more susceptible to dental caries due to weaker enamel properties and increased sensitivity during brushing. Research indicates that individuals with (MIH) experience higher rates of dental caries and require more frequent treatments. Therefore, it is crucial to implement a comprehensive preventive strategy as soon as lesions are detected on erupting first permanent molars. (MIH) can be categorized by the severity and extent of lesions, with three main degrees: mild, moderate, and severe. The mild form is characterized by opaque white discolorations of the enamel. Moderate cases show more significant discolorations, varying from yellow to brown. In severe cases, there is not only discoloration but also a marked loss of hard tissue, resulting in cavities or enamel fractures.

A systematic review done recommended the use of fissure sealants for mild cases of (MIH) in which first permanent molars do not exhibit posteruptive breakdown (PEB) and highlighted that Resin-based sealants are the most frequently utilized materials for this purpose.

creation of pre-reacted glass ionomer (PRG) filler technology in 1999 , which involves dispersing fluoroaluminosilicate glass particles that have already reacted with polyacrylic acid into resin. Building on this, a new hybrid material known as giomer was introduced, utilizing a bioactive surface pre-reacted glass (S-PRG) filler that merges the benefits of resin composites with those of glass ionomer cements Current evidence suggests that Phosphoric acid etching is the preferred method for sealing pits and fissures as it increases the retention rates. However, more high-quality multicenter randomized controlled trials are needed to explore the relationship between clinical effectiveness, retention rates especially in molars affected by (MIH) sealed by giomer-based fissure sealant preceded by etching using phosphoric acid etchant.

The benefits of this study to the participants:

1. Prevention of Complications: Early intervention can help prevent further enamel degradation and associated complications, e.g., Caries.
2. Improved Patient Comfort: Addressing hypersensitivity and pain early can enhance patient comfort.
3. Cost-Effectiveness: Preventive measures and early treatments can reduce overall treatment costs.

The benefits of this study to the clinicians:

1. Easier Management: Treating (MIH) when the condition is less severe allows for simpler and less invasive procedures.
2. Offering good alternative solutions for mild (MIH).

The benefits of this study to the population:

• Education Opportunities: Early diagnosis and treatment provide an opportunity for dentists to educate patients and families about oral health and the importance of regular dental visits and help them having better quality of life and prevent complications of untreated (MIH).

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 6-14 years who are diagnosed with mild (MIH) according to European Academy of Pediatric Dentistry (EAPD) criteria which includes demarcated enamel opacities (white, creamy, or yellow to brownish), that may induce sensitivity to external stimuli without enamel breakdown.

  * Cooperative children.
  * Presenting at least one first permanent molar (FPMs) that were fully erupted and indicated for non-invasive fissure sealant.
  * Medically fit Children (ASA I).

Exclusion Criteria:

* Children have hypomineralized (FPMs) with post-eruptive breakdown, cavitated and non-cavitated carious lesions, restorations, or fixed orthodontic appliances.
* Enamel defects due to a condition other than (MIH).
* Parents are not willing to join.
* Molars that cannot be isolated using rubber dam.
* Uncooperative children.
* Medically unfit children (other than ASA I).

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Sealant retention: Visual and tactile examination using dental mirror and dental probe using Modified (USPHS). | at 3 month, at 6 month and at 12 month.

SECONDARY OUTCOMES:
Anatomic form: Using Modified (USPHS) Criteria Visual and tactile examination using dental mirror and dental probe (Beste Özgür et al,2022). | at 3 month, at 6 month and at12 month.
• Marginal adaptation: Using Modified (USPHS) Criteria visual and tactile examination using dental mirror and dental probe (Beste Özgür et al,2022). | at 3 month, at 6 month and at 12 month.
• Marginal discoloration: using Modified (USPHS) Criteria visual examination using dental mirror (Beste Özgür et al,2022). | at 3 month, at 6 month and at 12 month.
• Surface texture: using Modified (USPHS) Criteria visual and tactile examination using dental mirror and dental probe (Beste Özgür et al,2022). | at 3 month, at 6 month and at 12 month.
• Secondary caries: Using Modified (USPHS) Criteria visual and tactile examination using dental mirror and dental probe (Beste Özgür et al,2022). | at 3 month, at 6 month and at 12 month.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wright JT, Tampi MP, Graham L, Estrich C, Crall JJ, Fontana M, Gillette EJ, Novy BB, Dhar V, Donly K, Hewlett ER, Quinonez RB, Chaffin J, Crespin M, Iafolla T, Siegal MD, Carrasco-Labra A. Sealants for Preventing and Arresting Pit-and-fissure Occlusal Caries in Primary and Permanent Molars. Pediatr Dent. 2016;38(4):282-308. PMID 27557916
- [Background] Toumba KJ, Twetman S, Splieth C, Parnell C, van Loveren C, Lygidakis NAlpha. Guidelines on the use of fluoride for caries prevention in children: an updated EAPD policy document. Eur Arch Paediatr Dent. 2019 Dec;20(6):507-516. doi: 10.1007/s40368-019-00464-2. Epub 2019 Nov 8. PMID 31631242
- [Background] Somani C, Taylor GD, Garot E, Rouas P, Lygidakis NA, Wong FSL. An update of treatment modalities in children and adolescents with teeth affected by molar incisor hypomineralisation (MIH): a systematic review. Eur Arch Paediatr Dent. 2022 Feb;23(1):39-64. doi: 10.1007/s40368-021-00635-0. Epub 2021 Jun 10. PMID 34110615
- [Background] 21. Singh D, Malik M, Mathur S. Comparative evaluation of clinical performance of giomer based and hydrophilic resin based pit and fissure sealant in primary molars: a split mouth clinical trial. J Pharm Negat Results. 2022;1883-9. 10.47750/pnr.2022.13.S04.229.
- [Background] 20. Ratnaditya A, Kumar M, Sai SAJ, Zabirunnisa M, Kandregula CR, Kopuri R. Clinical evaluation of Retention in Hydrophobic and Hydrophillic pit and fissure Sealants-A Two Year Follow-Up study. J Young Pharmacists. 2015. 10.5530/jyp.2015.3.6.
- [Background] Penha KJS, Roma FRVO, Filho EMM, Ribeiro CCC, Firoozmand LM. Bioactive self-etching sealant on newly erupted molars: A split-mouth clinical trial. J Dent. 2021 Dec;115:103857. doi: 10.1016/j.jdent.2021.103857. Epub 2021 Oct 24. PMID 34699954
- [Background] Ozgur B, Kargin ST, Olmez MS. Clinical evaluation of giomer- and resin-based fissure sealants on permanent molars affected by molar-incisor hypomineralization: a randomized clinical trial. BMC Oral Health. 2022 Jul 5;22(1):275. doi: 10.1186/s12903-022-02298-9. PMID 35790955
- [Background] Ntaoutidou S, Arhakis A, Tolidis K, Kotsanos N. Clinical evaluation of a surface pre-reacted glass (S-PRG) filler-containing dental sealant placed with a self-etching primer/adhesive. Eur Arch Paediatr Dent. 2018 Dec;19(6):431-437. doi: 10.1007/s40368-018-0379-z. Epub 2018 Oct 16. PMID 30328064
- [Background] Mohapatra S, Prabakar J, Indiran MA, Kumar RP, Sakthi DS. Comparison and Evaluation of the Retention, Cariostatic Effect, and Discoloration of Conventional Clinpro 3M ESPE and Hydrophilic Ultraseal XT Hydro among 12-15-year-old Schoolchildren for a Period of 6 Months: A Single-blind Randomized Clinical Trial. Int J Clin Pediatr Dent. 2020 Nov-Dec;13(6):688-693. doi: 10.5005/jp-journals-10005-1859. PMID 33976497
- [Background] Lopes LB, Machado V, Mascarenhas P, Mendes JJ, Botelho J. The prevalence of molar-incisor hypomineralization: a systematic review and meta-analysis. Sci Rep. 2021 Nov 17;11(1):22405. doi: 10.1038/s41598-021-01541-7. PMID 34789780
- [Background] Jorge RC, Dos Papoula GorniReis P, Maranon-Vasquez GA, Masterson D, Cople Maia L, Mendes Soviero V. Are yellow-brownish opacities in hypomineralized teeth more prone to breakage than white-creamy ones? A systematic review. Clin Oral Investig. 2022 Sep;26(9):5795-5808. doi: 10.1007/s00784-022-04536-4. Epub 2022 May 14. PMID 35568765
- [Background] Inchingolo AM, Inchingolo AD, Viapiano F, Ciocia AM, Ferrara I, Netti A, Dipalma G, Palermo A, Inchingolo F. Treatment Approaches to Molar Incisor Hypomineralization: A Systematic Review. J Clin Med. 2023 Nov 20;12(22):7194. doi: 10.3390/jcm12227194. PMID 38002806
- [Background] Hjertberg E, Hajdarevic A, Jalevik B. Desensitization treatment in MIH-affected teeth: a systematic review. Eur Arch Paediatr Dent. 2025 Feb;26(1):17-29. doi: 10.1007/s40368-024-00934-2. Epub 2024 Aug 13. PMID 39136874
- [Background] Hassan AM, Mohammed SG. Effectiveness of Seven Types of Sealants: Retention after One Year. Int J Clin Pediatr Dent. 2019 Mar-Apr;12(2):96-100. doi: 10.5005/jp-journals-10005-1600. PMID 31571779
- [Background] Lygidakis NA, Garot E, Somani C, Taylor GD, Rouas P, Wong FSL. Best clinical practice guidance for clinicians dealing with children presenting with molar-incisor-hypomineralisation (MIH): an updated European Academy of Paediatric Dentistry policy document. Eur Arch Paediatr Dent. 2022 Feb;23(1):3-21. doi: 10.1007/s40368-021-00668-5. Epub 2021 Oct 20. PMID 34669177
- [Background] Etman AM, Aboubakr RM, Alkhadragy D. Prevalence and predictors of molar-incisor hypomineralization among Egyptian children: a cross-sectional study. Eur Oral Res. 2024 Sep 5;58(3):120-126. doi: 10.26650/eor.20241394207. PMID 39588477
- [Background] Dimopoulou E, Baysan A. Effect of topical applications containing surface pre-reacted glass-ionomer filler on dental hard tissues-A systematic review. J Dent. 2024 Aug;147:104904. doi: 10.1016/j.jdent.2024.104904. Epub 2024 Mar 3. PMID 38442802
- [Background] 5. Comparative Evaluation Of Clinical Performance Of Giomer Based And Hydrophilic Resin Based Pit And Fissure Sealant In Primary Molars: A Split Mouth Clinical Trial" (2022) Journal of Pharmaceutical Negative Results, pp. 1883-1889
- [Background] Ciucchi P, Neuhaus KW, Emerich M, Peutzfeldt A, Lussi A. Evaluation of different types of enamel conditioning before application of a fissure sealant. Lasers Med Sci. 2015 Jan;30(1):1-9. doi: 10.1007/s10103-013-1333-2. Epub 2013 May 1. PMID 23636296
- [Background] AlGhannam MI, AlAbbas MS, AlJishi JA, AlRuwaili MA, AlHumaid J, Ibrahim MS. Remineralizing Effects of Resin-Based Dental Sealants: A Systematic Review of In Vitro Studies. Polymers (Basel). 2022 Feb 17;14(4):779. doi: 10.3390/polym14040779. PMID 35215692
- [Background] Almulhim B. Molar and Incisor Hypomineralization. JNMA J Nepal Med Assoc. 2021 Mar 31;59(235):295-302. doi: 10.31729/jnma.6343. PMID 34506432
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34669177/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39136874/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35568765/